CLINICAL TRIAL: NCT04826575
Title: High Intensity Respiratory Muscle Training as a Pre-habilitation in Lung Surgery
Brief Title: Pre-habilitation in Lung Surgery Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Brno University Hospital (Other); Palacky University (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, Ivan Cundrle M.D., Ph.D., St. Anne's University Hospital Brno, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NU21-06-00086
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer; Post-Op Complication
Keywords: cardiopulmonary exercise testing; VE/VCO2; PETCO2
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to control and intervention (pre-habilitation) group
Who Masked: Care Provider, Investigator
Masking Description: Caretaking provider and investigators gathering data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No intervention will be done in this group.
- Pre-Habilitation (Experimental): Two weeks of high intensity respiratory muscle training, optional smoking cessation and psychological support.
  Interventions: Other: High intensity inspiratory and expiratory muscle training

INTERVENTIONS:
Other: High intensity inspiratory and expiratory muscle training — Inspiratory Muscle Training will be performed using the Threshold inspiratory muscle trainer device (Threshold IMT®, Philips Respironics, Inc., Murrysville, PA, USA).
  Expiratory muscle training (EMT) will be performed using the Threshold positive expiratory pressure device (Threshold PEP®, Philips Respironics, Inc., Murrysville, PA, USA) or Expiratory Muscle Strength Trainer EMST 150TM (Aspire Products), depending on the initial MEP.
  Patients will train 2 times a day, 7 days per week, for 2 weeks.
  Arms: Pre-Habilitation

SUMMARY:
We hypothesize that high intensity respiratory muscle training will improve ventilatory efficiency (VE/VCO2 slope) and will be associated with decreased PPC, decreased mortality and better quality of life in lung resection candidates. Accordingly, the aim of this study will be to compare rest and exercise ventilation and gas exchange parameters as well as postoperative complications, quality of life and mortality in patients who undergo high intensity respiratory muscle training compared to patients who receive the usual standard of care.

DETAILED DESCRIPTION:
Lung resection surgery is the major curative option for lung cancer. Therefore, it is alarming that up to 37% of suitable patients are considered inoperable because of lung function impairment and those suitable for operation still carry a significant risk of especially postoperative pulmonary complications (PPC) development and increased mortality. Several predictors of postoperative morbidity and mortality have been identified. However, most of the factors are not easily modifiable before surgery. Ventilatory efficiency for carbon dioxide (VE/VCO2 slope) is an exercise parameter that has been shown to predict respiratory complications and mortality of lung resection candidates and to be superior to peak oxygen uptake (peak VO2). Importantly, in contrast to most previously established PPC risk factors, VE/VCO2 slope and peak VO2 may be therapeutically improved by physical and/or respiratory muscle training (e.g. by prehabilitation) and may thereby enable preoperative patient optimization. In thoracic surgery patients, trials looking at improvement of exercise capacity and PPC development give conflicting results, probably because of huge heterogeneity in terms of type, intensity and the length of pre-habilitation program. However, it seems that inclusion of only selected patients that may benefit from pre-habilitation (high risk patients), using VE/VCO2 slope and not peak VO2 to define the high risk patients and using interventions that could effectively improve VE/VCO2 slope (like the inspiratory and expiratory muscle training) is crucial and may be the key to lowering of postoperative pulmonary complications. Therefore, we hypothesize that high intensity respiratory muscle training will improve ventilatory efficiency (VE/VCO2 slope) and will be associated with decreased PPC, decreased mortality and better quality of life in lung resection candidates.

ELIGIBILITY:
Inclusion Criteria:

* ventilatory efficiency (VE/VCO2) ≥ 33

Exclusion Criteria:

* contraindication for lung resection (e.g. inoperable tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pulmonary complications | from the first 30 post-operative days or from the hospital stay
  Post-operative pulmonary complications
Post-operative cardiovascular complications | from the first 30 post-operative days or from the hospital stay
  Post-operative cardiovascular complications

SECONDARY OUTCOMES:
Hospital length of stay | from the first 30 post-operative days or from the hospital stay
  duration of hospital length of stay
Intensive care unit length of stay | from the first 30 post-operative days or from the hospital stay
  duration of intensive care unit length of stay
Chest drainage | from the first 30 post-operative days or from the hospital stay
  Duration of chest drainage

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, M.D., Ph.D., Principal Investigator — St. Anne's University Hospital in Brno
Locations (3):
- Czechia (3):
  - University Hospital Brno, Brno, Czech Republic
  - St. Anne's University Hospital, Brno, Czech Republic
  - Palacky University Olomouc, Olomouc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Lorente D, Navarro-Ripoll R, Guzman R, Moises J, Gimeno E, Boada M, Molins L. Prehabilitation in thoracic surgery. J Thorac Dis. 2018 Aug;10(Suppl 22):S2593-S2600. doi: 10.21037/jtd.2018.08.18. PMID 30345096
- [Background] Baser S, Shannon VR, Eapen GA, Jimenez CA, Onn A, Keus L, Lin E, Morice RC. Pulmonary dysfunction as a major cause of inoperability among patients with non-small-cell lung cancer. Clin Lung Cancer. 2006 Mar;7(5):344-9. doi: 10.3816/CLC.2006.n.017. PMID 16640807
- [Background] Agostini P, Cieslik H, Rathinam S, Bishay E, Kalkat MS, Rajesh PB, Steyn RS, Singh S, Naidu B. Postoperative pulmonary complications following thoracic surgery: are there any modifiable risk factors? Thorax. 2010 Sep;65(9):815-8. doi: 10.1136/thx.2009.123083. PMID 20805178
- [Background] Brunelli A, Varela G, Refai M, Jimenez MF, Pompili C, Sabbatini A, Aranda JL. A scoring system to predict the risk of prolonged air leak after lobectomy. Ann Thorac Surg. 2010 Jul;90(1):204-9. doi: 10.1016/j.athoracsur.2010.02.054. PMID 20609776
- [Background] Stanzani F, Paisani Dde M, Oliveira Ad, Souza RC, Perfeito JA, Faresin SM. Morbidity, mortality, and categorization of the risk of perioperative complications in lung cancer patients. J Bras Pneumol. 2014 Jan-Feb;40(1):21-9. doi: 10.1590/S1806-37132014000100004. PMID 24626266
- [Background] Brunelli A, Belardinelli R, Pompili C, Xiume F, Refai M, Salati M, Sabbatini A. Minute ventilation-to-carbon dioxide output (VE/VCO2) slope is the strongest predictor of respiratory complications and death after pulmonary resection. Ann Thorac Surg. 2012 Jun;93(6):1802-6. doi: 10.1016/j.athoracsur.2012.03.022. Epub 2012 May 4. PMID 22560968
- [Background] Torchio R, Guglielmo M, Giardino R, Ardissone F, Ciacco C, Gulotta C, Veljkovic A, Bugiani M. Exercise ventilatory inefficiency and mortality in patients with chronic obstructive pulmonary disease undergoing surgery for non-small-cell lung cancer. Eur J Cardiothorac Surg. 2010 Jul;38(1):14-9. doi: 10.1016/j.ejcts.2010.01.032. Epub 2010 Mar 30. PMID 20356758
- [Background] Fu TC, Wang CH, Lin PS, Hsu CC, Cherng WJ, Huang SC, Liu MH, Chiang CL, Wang JS. Aerobic interval training improves oxygen uptake efficiency by enhancing cerebral and muscular hemodynamics in patients with heart failure. Int J Cardiol. 2013 Jul 15;167(1):41-50. doi: 10.1016/j.ijcard.2011.11.086. Epub 2011 Dec 22. PMID 22197120
- [Background] Tucker WJ, Lijauco CC, Hearon CM Jr, Angadi SS, Nelson MD, Sarma S, Nanayakkara S, La Gerche A, Haykowsky MJ. Mechanisms of the Improvement in Peak VO2 With Exercise Training in Heart Failure With Reduced or Preserved Ejection Fraction. Heart Lung Circ. 2018 Jan;27(1):9-21. doi: 10.1016/j.hlc.2017.07.002. Epub 2017 Aug 4. PMID 28870770
- [Background] Kasahara Y, Izawa KP, Watanabe S, Osada N, Omiya K. The Relation of Respiratory Muscle Strength to Disease Severity and Abnormal Ventilation During Exercise in Chronic Heart Failure Patients. Res Cardiovasc Med. 2015 Sep 15;4(4):e28944. doi: 10.5812/cardiovascmed.28944. eCollection 2015 Nov. PMID 26528451
- [Derived] Filakovszky A, Brat K, Tschoellitsch T, Bartos S, Mazur A, Meier J, Olson L, Cundrle I. Cardiopulmonary exercise testing before lung resection surgery: still indicated? Evaluating predictive utility using machine learning. Thorax. 2025 Oct 2:thorax-2024-221485. doi: 10.1136/thorax-2024-221485. Online ahead of print. PMID 41043965